CLINICAL TRIAL: NCT05608603
Title: Observational Cohort Prospective Study of Diagnostics of Coronavirus Disease 2019 Cardiovascular Complications Using Remote Electrocardiogram Monitoring and Pulse Wave
Brief Title: Diagnostics of Coronavirus Disease 2019 Cardiovascular Complications
Status: Enrolling by invitation | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 12211
Record Dates: First submitted 2022-11-05; First posted 2022-11-08 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Endothelial Function; Diastolic Dysfunction; Oxygen Consumption; Quality of Life; Exercise Tolerance
Keywords: COVID-19; markers of endothelial function; diastolic dysfunction; oxygen consumption; flow mediated dilatation; proton mass spectrometry; remote ECG monitoring; pulse vawe
MeSH Terms: conditions — COVID-19 | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3 months postcovid patients: Included 100 patients, aged 18-80 years old, at 3 months after infection COVID-19.
  Intervention: cardiorespiratory stress test to determine the patient's oxygen consumption; electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark"; the analysis of exhaled air will be performed using the Compact PTR-MS proton mass spectrometer manufactured by Ionicon (Austria).
  Interventions: Diagnostic Test: Portable cardiac monitor "CardioQvark"; Diagnostic Test: Cardiorespiratory stress test; Diagnostic Test: Analysis of exhaled air using the Compact PTR-MS proton mass spectrometer
- 9 months postcovid patients: Included the same 100 patients, aged 18-80 years old, at 9 months after infection COVID-19.
  Intervention: cardiorespiratory stress test to determine the patient's oxygen consumption; electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark"; the analysis of exhaled air will be performed using the Compact PTR-MS proton mass spectrometer manufactured by Ionicon (Austria).
  Interventions: Diagnostic Test: Portable cardiac monitor "CardioQvark"; Diagnostic Test: Cardiorespiratory stress test; Diagnostic Test: Analysis of exhaled air using the Compact PTR-MS proton mass spectrometer

INTERVENTIONS:
Diagnostic Test: Portable cardiac monitor "CardioQvark" — Record an electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark" (Russia, LLC "L Card" , RU No. RZN 2019/8124 dated February 15, 2019) once. Devices automatically transfer data to the A&D Connect app paired with it (link). When transferring data, they are completely protected. The data obtained using the application must be sent to the specialists of the research group in a depersonalized form.
  Other Names: Electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark"
Diagnostic Test: Cardiorespiratory stress test — Cardiorespiratory stress testing with gas analysis using the Quark CPET diagnostic system (COSMED, Italy). The study protocol will consist of 4 phases: rest, warm-up, exercise and recovery. During the load phase, a ramp protocol will be used with a stepped load from 10 to 25 W/min. The increase in power will be calculated individually before the start of the study so that the test lasts 8-12 minutes until complete muscle failure.
Diagnostic Test: Analysis of exhaled air using the Compact PTR-MS proton mass spectrometer — The analysis of exhaled air will be performed using the Compact PTR-MS proton mass spectrometer manufactured by Ionicon (Austria)

SUMMARY:
Aim of this prospective, observational, multi-centered, randomized study is to detect cardiovascular complications in patients after coronavirus infection.

The study will include 100 patients who underwent confirmed by laboratory tests COVID-19 infection (polymerase chain reaction (PCR) testing, enzyme-linked immunosorbent assay (positive result at least 1 time)) 1-3 months ago with the degree of lung lesion more than 25%, who were admitted to the University Clinical Hospital No. 4 of I.M. Sechenov First Moscow State Medical University.

The study consists of 4 periods:

1. Screening for up to 6 months.
2. Inclusion in the study, undergoing of identical laboratory and instrumental testing.
3. Re-examination of patients. After 6 months from the initial examination (9 months after discharge from the infectious diseases department), patients will be re-examined.

4 Determination of end points, statistical data processing.

Estimated result of the study is to confirm or refute the hypothesis:

1. As a result of the analysis of ECG and pulse wave data and comparison with echocardiography data, identify cardiovascular complications of COVID-19 infection.
2. To determine the diagnostic significance of pulse wave parameters for assessing cardiovascular complications in patients with a history of COVID-19 infection (sensitivity, specificity, positive and negative predictive value).
3. Identify correlations between pulse wave parameters and biochemical markers of endothelial dysfunction (endothelin-1).
4. As a result of the analysis of exhaled air by the proton mass spectrometry, to identify markers of cardiovascular complications in patients after COVID-19 infection.
5. As a result of a cardiorespiratory stress test, determine the respiratory and cardiovascular causes of dyspnea, exercise tolerance of patients after infection with COVID-19.

DETAILED DESCRIPTION:
Aim of this prospective, observational, multi-centered, randomized study is to detect cardiovascular complications in patients after coronavirus infection.

The study will include 100 patients who underwent confirmed by laboratory tests Coronavirus Disease 2019 (COVID-19) infection (polymerase chain reaction (PCR) testing, enzyme-linked immunosorbent assay (positive result at least 1 time)) 1-3 months ago with the degree of lung lesion more than 25%, who were admitted to the University Clinical Hospital No. 4 of I.M. Sechenov First Moscow State Medical University.

The study consists of 4 periods:

1. Screening for up to 6 months. Performed by a pulmonologist. Patients meeting the inclusion criteria are selected.
2. Inclusion in the study. If the patient meets the inclusion criteria, a discussion about the nature of the study is held with the patient. Further, consent to participate in the study and to process personal data is obtained. After, the epicrisis from the COVID-19 infectious diseases department is analyzed.

   Patients are provided with medical care in accordance with the standards approved by the Ministry of Health of the Russian Federation, and local acts of the institution in which the study is carried out.

   Patients eligible for inclusion will undergo the following investigations:
   * Anamnesis and complaints collection; physical examination;
   * Assessment of the quality of life and psycho-emotional status using the Short Form-36 (SF36) and Hospital Anxiety and Depression Scale (HADS) questionnaires, as well as the six-minute walk test;
   * General and biochemical blood tests , urine analysis, , determination of biochemical markers of endothelial dysfunction (endothelin-1) in the blood;
   * Electrocardiography, a flow mediated dilatation procedure for endothelial function assessment, transthoracic echocardiography to identify the structural and functional features of the myocardium, spiroergometry to determine the patient's oxygen consumption.
   * Electrocardiogram (ECG) in one lead with an assessment of the pulse wave using a portable cardiac monitor "CardioQvark"
   * The analysis of exhaled air will be performed using the Compact proton mass spectrometer (PTR-MS) manufactured by Ionicon (Austria).
3. Re-examination of patients. After 6 months from the initial examination (9 months after discharge from the infectious diseases department), patients will be re-examined, In the interval between the initial and repeated examinations, the condition of all patients will be monitored, for this it is expected to make phone calls, the frequency of 1 time per month.

4 Determination of end points, statistical data processing. The statistical processing will be performed using the Python Software Foundation version 3.8 for Windows (Delaware, USA).

Estimated result of the study is to confirm or refute the hypothesis:

1. As a result of the analysis of ECG and pulse wave data and comparison with echocardiography data, identify cardiovascular complications of COVID-19 infection.
2. To determine the diagnostic significance of pulse wave parameters for assessing cardiovascular complications in patients with a history of COVID-19 infection (sensitivity, specificity, positive and negative predictive value).
3. Identify correlations between pulse wave parameters and biochemical markers of endothelial dysfunction (endothelin-1).
4. As a result of the analysis of exhaled air by the proton mass spectrometry, to identify markers of cardiovascular complications in patients after COVID-19 infection.
5. As a result of a cardiorespiratory stress test, determine the respiratory and cardiovascular causes of dyspnea, exercise tolerance of patients after infection with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study;
2. Age 18 and over;
3. Male and female;
4. COVID-19 infection confirmed by laboratory tests (polymerase chain reaction testing, enzyme-linked immunosorbent assay (positive result at least 1 time) with a CT degree more that 25% of lung lesion.
5. No more than 3 months after discharge from infectious department

Non-inclusion criteria:

1. Unable to sign informed consent;
2. Mental illness (severe dementia, schizophrenia, severe depression, manic-depressive psychosis);
3. Acute coronary syndrome, acute cerebrovascular accident, pulmonary embolism within the last 3 months;
4. Oncology;
5. Diseases and conditions that can change the ECG picture and complicate the analysis of the ECG (conduction disturbance, pacemaker);
6. Inability to use a heart monitor (congenital developmental anomalies, traumatic amputation of the upper limbs, essential tremor, Parkinson's disease);
7. Severe comorbidities with life expectancy less than 1 year.

Exclusion Criteria:

1. Refusal to further participation in the study;
2. Acute infectious diseases, tuberculosis
3. Oncology arising in the process of the study
4. Acute coronary syndrome, acute cerebrovascular accident, pulmonary embolism arising in the process of the study
5. Acute psychotic reactions arising in the process of the study;
6. Inability to use a heart monitor arising in the process of the study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consist all men and women from 18 to 80 age in a community according inclusion, non-inclusion, exclusion criteria
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in endothelin-1 in dynamics (compared with initial indicators) | In 9 months after the recovery from COVID-19
  This outcome will be assessed by taking blood samples from a peripheral vein
Changes in the diastolic function of the right and left ventricles (compared with initial indicators) | In 9 months after the recovery from COVID-19
  Transthoracic echocardiography (EchoCG) will be performed to assess the heart structure and function: unidimensional (M-mode), two-dimensional (B-mode) and Doppler.
  Diastolic function of the left ventricle will be assessed using pulse-wave, constant-wave, and tissue Doppler studies. Maximum velocity of early (E peak) and late (A peak) diastolic filling, E/A ratio, time of blood flow deceleration of early left ventricular diastolic filling (DT) will be determined at simultaneous recording of aortic and transmitral blood flow in constant-wave mode, left ventricular isovolumic relaxation time (IVRT) - interval from the end of aortic to the beginning of transmitral blood flow.
Change in ejection fraction (compared with initial indicators) | In 9 months after the recovery from COVID-19
  Transthoracic EchoCG will be performed to assess the heart structure and function: unidimensional (M-mode), two-dimensional (B-mode) and Doppler.
  Ejection fraction will be assessed according to BIPLANE, TAPSE.
Changes in the volumes of the heart cavities (compared with initial indicators) | In 9 months after the recovery from COVID-19
  Transthoracic EchoCG will be performed to assess the heart structure and function: unidimensional (M-mode), two-dimensional (B-mode) and Doppler.
Change in speed indicators on the heart valves (compared with initial indicators) | In 9 months after the recovery from COVID-19
  Transthoracic EchoCG will be performed to assess the heart structure and function: unidimensional (M-mode), two-dimensional (B-mode) and Doppler.
Change in mean and diastolic pressure of the pulmonary artery (compared with initial indicators) | In 9 months after the recovery from COVID-19
  Transthoracic EchoCG will be performed to assess the heart structure and function: unidimensional (M-mode), two-dimensional (B-mode) and Doppler.
Changes in the cardio-ankle vascular index and ankle-brachial index (compared with initial indicators) | In 9 months after the recovery from COVID-19
  Will be assessed by using pulse wave measurements in dynamics
Changes in the spectrum of volatile organic compounds in exhaled air in patients after COVID-19 infection over time (compared with initial indicators) | In 9 months after the recovery from COVID-19
  Will be assessed by using exhale air proton mass spectrometry in dynamics.
Change in oxygen pulse (VO2/HR) at the peak of the load | In 9 months after the recovery from COVID-19
  The spiroergometric test will be performed under continuous stepwise increasing load. The duration of each load step is 5 min; the initial load level is 25 W, followed by an increase in load at each step by the same amount. The results of the test will be used to evaluate the achievement of the maximum level of oxygen consumption (in l/min or ml/min/kg body weight) and the maximum achievement of the "oxygen pulse" on load.
Changes in ventilation parameters (tidal volume (Vt), minute ventilation (VE), Vt/FVC index (ratio of tidal volume to forced vital capacity), respiratory reserve (BR)) over time | In 9 months after the recovery from COVID-19
  The spiroergometric test will be performed under continuous stepwise increasing load. The duration of each load step is 5 min; the initial load level is 25 W, followed by an increase in load at each step by the same amount. The results of the test will be used to evaluate the achievement of the maximum level of oxygen consumption (in l/min or ml/min/kg body weight) and the maximum achievement of the "oxygen pulse" on load.
Changes in gas exchange parameters (end-expiratory partial pressure of exhaled carbon dioxide (PetCO2), ventilation equivalent for carbon dioxide (VE/VCO2), ventilation-perfusion ratio (Vd/Vt)) in dynamics | In 9 months after the recovery from COVID-19
  The spiroergometric test will be performed under continuous stepwise increasing load. The duration of each load step is 5 min; the initial load level is 25 W, followed by an increase in load at each step by the same amount. The results of the test will be used to evaluate the achievement of the maximum level of oxygen consumption (in l/min or ml/min/kg body weight) and the maximum achievement of the "oxygen pulse" on load.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Yu Kopylov, Professor, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University)ogy, Center "Digital biodesign and personalized healthcare"), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Prohibition of local ethics committee